CLINICAL TRIAL: NCT01561898
Title: A Long-Term Study of JNS007ER in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Medical Director, Janssen Pharmaceutical K.K., Japan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012628; JNS007ER-JPN-S32 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Results first posted 2012-09-10 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; JNS007ER; Paliperidone extended-release
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone extended-release (JNS007ER) (Experimental)
  Interventions: Drug: Paliperidone extended-release (JNS007ER)

INTERVENTIONS:
Drug: Paliperidone extended-release (JNS007ER) — Type= range, unit= mg, number= 3-12, form= tablet, route= oral use. JNS007ER within the range of 3, 6, 9 and 12 mg will be orally administered once daily for 48 weeks.

SUMMARY:
The purpose of this study is to assess the safety of JNS007ER 3-12 mg once daily in patients with schizophrenia over a long term period.

DETAILED DESCRIPTION:
This is a 48-week, multicenter, open-label (all people know the identity of the intervention), non-controlled, arbitrary-dose study. The patients included in this study are those who participated in the preceding double-blind (neither physician nor patient knows the treatment that the patient receives) comparative trial (study JNS007ER-JPN-S31) of JNS007ER and completed the study, or those who remained in the study up to the evaluation at 2 weeks and discontinued the study after that for insufficient treatment efficacy. The study will assess the safety of JNS007ER in the clinical recommended dose range in a long term treatment. The dosage will be started at 6 mg/day, and it can be increased or decreased 3 mg at a time depending on the patient's symptom within the range of 3 mg/day to 12 mg/day. For dose adjustments, the investigator will evaluate the psychiatric symptoms before defining the dose change.

Detailed Description: Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia
* Patients who have given their own consent in writing to participate in the study
* Patients untreated with antipsychotics within 28 days before the screening test
* Patients who have completed Study JNS007ER-JPN-S31, or those who continued the study at least up to the evaluation at 2 weeks and subsequently discontinued the study due to insufficient efficacy
* Patients participating in Study JNS007ER-JPN-S31 and whose ratio of treatment to the evaluation at 2 weeks is ≥75%

Exclusion Criteria:

* Patients diagnosed with a mental disease other than schizophrenia
* A total PANSS score > 120 at baseline
* Substance-related disorders
* Parkinson's disease complications
* Current or a past history of convulsive disease such as epilepsy
* Current or a past history of cerebrovascular accident
* Diabetes mellitus
* Significant hepatic or renal impairment
* Significant cardiovascular disorders
* Abnormal results of hematological examination, blood chemistry test and urinalysis at screening
* Pregnant women, breast-feeding mothers, and patients who wish pregnancy during the study period or those whose pregnancy test at screening was positive
* Contraindications to risperidone products
* Patients who discontinued Study JNS007ER-JPN-S31 due to an adverse event not related to the underlying disease
* Patients judged inadequate by the investigator to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study comprises patients who have participated in previous study JNS007ER-JPN-S31 (NCT00396565) and new patients. New patients were classified as group NO/PAL. Patients entering from study JNS007ER-JPN-S31 were classified according to their origin groups: placebo group (PLA/PAL), paliperidone group (PAL/PAL), and olanzapine group (OLZ/PAL).
Groups:
- NO/PAL Group: NO/PAL: group consisting of new patients. Treatment is started with paliperidone extended release (ER) 6 mg once daily, and the dose is appropriately increased or decreased within the range from 3mg to 12 mg.
- PLA/PAL Group: PLA/PAL: group of continuing patients from JNS007ER-JPN-S31 in which they belonged to the placebo group. Treatment is started with paliperidone extended release (ER) 6 mg once daily, and the dose is appropriately increased or decreased within the range from 3mg to 12 mg.
- PAL/PAL Group: PAL/PAL: group of continuing patients from JNS007ER-JPN-S31 in which they belonged to the paliperidone ER group. Treatment is started with paliperidone extended release (ER) 6 mg once daily, and the dose is appropriately increased or decreased within the range from 3mg to 12 mg.
- OLZ/PAL: OLZ/PAL: group of continuing patients from JNS007ER-JPN-S31 in which they belonged to the olanzapine group. Treatment is started with paliperidone extended release (ER) 6 mg once daily, and the dose is appropriately increased or decreased within the range from 3mg to 12 mg.
Period: Overall Study
Arm/Group | NO/PAL Group | PLA/PAL Group | PAL/PAL Group | OLZ/PAL
Started | 7 | 92 | 97 | 32
Completed | 5 | 51 | 53 | 12
Not Completed | 2 | 41 | 44 | 20
Not completed — Withdrawal by Subject | 0 | 8 | 12 | 5
Not completed — Lack of Efficacy | 0 | 8 | 10 | 5
Not completed — Worsening of complications | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 19 | 14 | 9
Not completed — Physician Decision | 1 | 5 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NO/PAL Group | PLA/PAL Group | PAL/PAL Group | OLZ/PAL | Total
Number analyzed (Participants) | 7 | 92 | 97 | 32 | 228
Age Continuous [Mean (Standard Deviation); unit: years] | 35.6 (14.8) | 46.6 (15.5) | 42.0 (14.1) | 46.3 (14.0) | 44.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 44 | 46 | 20 | 113
  Male | 4 | 48 | 51 | 12 | 115

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS)
Description: PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Time Frame: Baseline, Week 48
Population: Intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- NO/PAL: NO/PAL: group consisting of new patients. Treatment is started with paliperidone extended release (ER) 6 mg once daily, and the dose is appropriately increased or decreased within the range from 3mg to 12 mg.
Arm/Group | NO/PAL | PLA/PAL Group | PAL/PAL Group | OLZ/PAL
Number analyzed (Participants) | 7 | 92 | 97 | 32
scores on a scale | -13.4 (31.93) | -11.1 (20.84) | -17.2 (22.15) | 2.8 (20.67)

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S)
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients".
Time Frame: Baseline, Week 48
Population: Intent-to-treat (ITT) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NO/PAL | PLA/PAL Group | PAL/PAL Group | OLZ/PAL
Number analyzed (Participants) | 7 | 92 | 97 | 32
scores on a scale | -0.6 (1.27) | -0.6 (1.20) | -0.7 (1.24) | 0.1 (1.01)

3. Primary Outcome: Incidence of Adverse Events
Description: The incidence of adverse events was measured by the percentage of patients who presented one or more adverse events.
Time Frame: 48 weeks
Population: Intent-to-treat (ITT) population
Measure: Number; unit: percentage of patients
Groups:
- Entire Group: Treatment is started with paliperidone extended release (ER) 6 mg once daily, and the dose is appropriately increased or decreased within the range from 3mg to 12 mg.
Arm/Group | Entire Group
Number analyzed (Participants) | 228
percentage of patients | 97.4

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Entire Group
Serious Adverse Events (participants affected / at risk) | 10/228
Other Adverse Events (participants affected / at risk) | 222/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Group (N=228)
Schizophrenia (Psychiatric disorders) | 3
Pneumonia (Infections and infestations) | 2
Insomnia (Psychiatric disorders) | 1
Akathisia (Nervous system disorders) | 1
Pulmonary aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Multiple organ failure (General disorders) | 1
ECG corrected QT interval prolonged (Cardiac disorders) | 1
Overdose (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Group (N=228)
Blood prolactin increased (Investigations) | 91
Nasopharyngitis (Infections and infestations) | 77
Schizophrenia (Psychiatric disorders) | 69
Weight increased (General disorders) | 50
Extrapyramidal disorder (Nervous system disorders) | 39
Constipation (Gastrointestinal disorders) | 32
Blood triglycerides increased (Metabolism and nutrition disorders) | 23
Blood creatine phosphokinase increased (Metabolism and nutrition disorders) | 28
Insomnia (Psychiatric disorders) | 23
Eczema (Skin and subcutaneous tissue disorders) | 20
Dental caries (Gastrointestinal disorders) | 16
Headache (Nervous system disorders) | 15
Fever (General disorders) | 15
Diarrhea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 14
Abnormal hepatic function (Hepatobiliary disorders) | 14
Backache (Musculoskeletal and connective tissue disorders) | 13
Blood cholesterol increased (Metabolism and nutrition disorders) | 13
Abrasion (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.